CLINICAL TRIAL: NCT01049815
Title: A Randomized-controlled Trial Comparing the Efficacy of Two Phosphorous Binders, Renagel and Caltrate in Reducing the Rate of Progression of Femoral and Carotid IMT Thickening as Measured by B-mode Ultrasound in Dialysis Patients.
Brief Title: Sevelamer Hydrochloride and Femoral and Carotid Intima Media Thickness Progression in End Stage Renal Disease
Acronym: SUMMER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Wolfson Medical Center (Other Government); Genzyme, a Sanofi Company (Industry)
Responsible Party: Talia Weinstein MD PhD, Tel Aviv Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-285
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: End Stage Renal Disease; Hemodialysis; Intimal Media Thickness
Keywords: hemodialysis; intimal media thickness
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Sevelamer; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevelamer hydrochloride (Experimental)
  Interventions: Drug: sevelamer hydrochloride
- Calcium carbonate (Active Comparator)
  Interventions: Drug: Calcium Carbonate

INTERVENTIONS:
Drug: sevelamer hydrochloride — 800-3200 mg with each meal
  Other Names: Renagel
  Arms: Sevelamer hydrochloride
Drug: Calcium Carbonate — 600 mg with each meal, up to 1800 mg a day
  Other Names: Caltrate, Calcimor
  Arms: Calcium carbonate

SUMMARY:
Aims of the multi-center, randomized, treatment-controlled clinical trial are to compare the efficacy of sevelamer hydrochloride to calcium-containing phosphorus binders in reducing the rate of progression of femoral and carotid intimal media thickness (IMT) thickening as measured by B-mode ultrasound in stable maintenance hemodialysis (HD) patients.

DETAILED DESCRIPTION:
Serum phosphorus (P) is frequently elevated in HD patients. Serum P stimulates PTH synthesis and is associated with secondary hyperparathyroidism. Use of calcium(Ca)-containing phosphorus-binders is an exogenous source of Ca that can elevate the CaxP product. In HD patients, an ultrasonographically-demonstrated increase in intima media thickness of the carotid artery has been associated with elevated serum P levels.Peripheral arterial vascular disease (PVD) accounts for significant mortality and morbidity in HD patients.

The aim of this study is to compare the efficacy of sevelamer hydrochloride to calcium-containing phosphorus binders in reducing the rate of progression of femoral and carotid intimal media thickness (IMT) thickening as measured by B-mode ultrasound in stable HD patients.

Subject randomization numbers was provided by the Epidemiology and Research Unit, E. Wolfson Medical Center, Holon, Israel. After meeting all inclusion criteria, subjects were randomized to one of two treatment groups: Renagel or calcium carbonate. Prior to receiving treatment, baseline femoral and carotid IMT were measured, medical and pharmaceutical history was documented, nutrition assessment was undertaken and midweek blood chemistry and blood count were measured. No change in patient medication prescription was required during this study, with the exception of phosphorus binders. All other concomitant medications were continued. During the year of the study, routine monthly blood tests were obtained for chemistry, blood count, and PTH was measured once every 4 months.

After a year of treatment, femoral and carotid IMT were measured again, midweek blood chemistry and blood count were measured.

ELIGIBILITY:
Inclusion Criteria:

* HD Patients aged 40-75 years inclusive if they received HD treatment three times each week for not less than three months, and if they had not been treated with sevelamer hydrochloride. Patients of both genders, without regard to diabetes status, history of CVD or underlying renal disease were eligible.

Exclusion Criteria:

* Patients receiving treatment with sevelamer hydrochloride were not eligible for study participation. Additionally, patients were excluded if they had active liver disease, known sensitivity to either sevelamer hydrochloride or calcum carbonate or if their participation in the study was deemed in any way detrimental or unwarranted by the patient's treating physician.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2005-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Increase in carotid and femoral IMT as measured using B-mode ultrasonography | 1 year

SECONDARY OUTCOMES:
Clinically evident PVD in a previously unaffected limb confirmed by doppler or duplex ultrasonography. Also, serum P, serum Ca, PTH and % of treatment group compliant with the revised treatment goals . | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Talia Weinstein, MD PhD, Principal Investigator — Tel Aviv Medical Center; Mona Boaz, PhD, Principal Investigator — Edith Wolfson Medical Center
Locations (2):
- Israel (2):
  - Edith Wolfson Medical Center, Holon
  - Tel Aviv Medical Center, Tel Aviv

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086